CLINICAL TRIAL: NCT02104375
Title: The Effects of L-Citrulline Supplementation on Vascular and Cardiac Autonomic Responses to Cold Pressor Test Concurrent With Postexercise Muscle Ischemia
Brief Title: L-citrulline Supplementation, Cold Exposure, & Post-Exercise Muscle Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2013.11742
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: wave reflection; augmentation Index; heart rate variability; arterial stiffness
MeSH Terms: conditions — Hypertension | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-citrulline (Experimental): L-citrulline (6 g/day for 2 weeks)
  Interventions: Dietary Supplement: L-citrulline
- Maltodextrin (Placebo Comparator): 6g/day of placebo (maltodextrin)
  Interventions: Dietary Supplement: L-citrulline

INTERVENTIONS:
Dietary Supplement: L-citrulline — 2 weeks of L-citrulline supplementation (6g/day).
  Other Names: 2 weeks of L-citrulline supplementation (6g/day).

SUMMARY:
Cardiovascular disease (CVD) continues to be the major cause of morbidity and mortality in western countries. It has been shown that CVD events are known to be higher in the winter than in the summer. Low environmental temperatures may induce increased cardiovascular stress resulting in cold-induced hypertension (CIH), the leading risk factor for CVD events. Similar to whole-body cold exposure, the cold pressor test (CPT), an external local cold stimulus, has been used for evaluation of cardiovascular and hemodynamic reactivity to sympathetic stimulation. It has been shown that brachial blood pressure (BP), pressure pulse wave reflection, aortic BP, heart rate (HR), and arterial stiffness are increased during CPT. However, the physiologic mechanisms for the cardiovascular complications related to low temperatures are not completely clear.

Isometric-handgrip (IHG) exercise has been used as a tool for assessing cardiovascular autonomic control by a maneuver defined as post-exercise muscle ischemia (PEMI). PEMI induces exercise pressor reflex (metaboreflex) by trapping metabolites in the previous active muscle at the cessation of exercise. During PEMI, the accumulation of contraction-derived metabolites induces sympathetic mediated vascular stimulation and an increased BP, whereas the HR fully recovers. This suggests that the fall in HR is evoked by an increase in parasympathetic activity which overpowers the sympathetic activation. Implication of IHG exercise followed by PEMI provides important clinical information because impaired autonomic and cardiovascular functions are associated with cardiovascular events.

Recently, oral supplementation with the amino acid L-citrulline (L-cit) has been proposed as a possible adjunct treatment for hypertension and arterial stiffness. L-cit is known to enhance the bioavailability of L-arginine (L-arg), the endothelial substrate for nitric oxide (NO) production. Cold exposure might include a temperature-dependent inhibition of endothelial NO synthase (eNOS), the enzyme that produces NO from the amino acid L-arg and may trigger various types of CVD. It has been shown that L-cit supplementation has effectively attenuated the CIH response during cold pressor test. Thus, L-cit supplementation may be effective to reduce the cardiovascular responses associated with cold exposure and the exercise pressor reflex imposed by PEMI. Therefore, the proposed study is important for the following reasons: (1) the results of his study will add to our understanding regarding the cardiovascular and autonomic mechanisms associated with exercise and cold exposure; (2) the results of this study will contribute to the development of an adjunct therapy for the prevention of cardiovascular adverse events that are particularly increased during stress such as cold exposure and exercise.

DETAILED DESCRIPTION:
Specific Aims

AIM 1: To determine the acute effects of the exercise pressor response imposed by PEMI with and without CPT on hemodynamics and cardiac autonomic regulation in health overweight/obese men.

AIM 2: To examine the effects of a 14-day course of L-cit supplementation on arterial stiffness, aortic hemodynamics, and autonomic regulation at rest and during conditions characterized by increased sympathetic activity (IHG, PEMI, and PEMI concurrent with CPT).

Research Hypotheses

Hypothesis 1: There will be greater increases in peripheral and central BP, arterial stiffness, wave reflection, and cardiac sympathetic activity during PEMI concurrent with CPT than during PEMI alone.

Hypothesis 2: 14 days of L-cit supplementation will attenuate peripheral and central BP, wave reflection, arterial stiffness, and cardiac sympathetic activity responses during IHG exercise, PEMI, and PEMI concurrent with CPT compared with placebo (PL) supplementation.

Description of the study

A total of twenty male young adults (18-35 years) with overweight or obesity [body mass index (BMI) >25 and <40 kg/m2] will be enrolled in this study. All of the subjects will be nonsmokers, no L-cit or L-arg users or regular exercisers (defined as more than 120 min per week) at least 6 months before the study begins. Subjects will be asked to maintain their diet and exercise habits during the study period.

Study design:

After completion of initial screening, cardiovascular and autonomic function of eligible subjects will be evaluated in a quiet temperature-controlled room (22-24°C). After baseline measurement, in a cross-over design fashion, subjects will be randomized to either Placebo group (Maltodextrin) or L-citrulline group for the first 14 days of the study that will be followed by a 14 day washout period and then will be crossed over to their next treatment. Cardiovascular function will be evaluated at baseline and after 14 days of the first and the second treatment. Measurements will be conducted in the morning after at least 8 hours of an overnight fast in order to avoid potential diurnal variations in BP and vascular reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Blood pressure lower than 140/90mmHg
* Age 18 to 35 years
* BMI 25-39 kg/m2

Exclusion Criteria:

* Blood Pressure >160/100 mmHg
* Asthma
* Glaucoma
* Herpes simplex
* Uncontrolled diabetes
* Neurological disease
* Cardiovascular disease
* Inflammatory disease
* Kidney disease
* Hormone replacement therapy (HRT)
* Amino acid/vitamin supplementation\
* Corticosteroids or non-steroidal anti-inflammatory drugs
* Any drug known to affect BP or heart rate
* Glycemic control drugs
* Lipids reducing drugs
* Participants should not consume > 12 alcoholic drink/week
* Smokers
* Regular Exercisers (>1.5 hour/week).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 6 weeks
  By measuring brachial and central (aortic and carotid) BP at rest and during physiological stress (cold pressor test, post-exercise muscle ischemia, and handgrip test)

SECONDARY OUTCOMES:
Arterial Stiffness | 6 weeks
  By measuring brachial-ankle pulse wave velocity at rest and during physiological stress (cold pressor test, post-exercise muscle ischemia, and handgrip test)

OTHER OUTCOMES:
Autonomic control of heart rate | 6 weeks
  By measuring heart rate variability at rest and during physiological stress.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, Principal Investigator — Florida State University
Locations (1):
- FSU College of Human Sciences, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Kalfon R, Campbell J, Alvarez-Alvarado S, Figueroa A. Aortic Hemodynamics and Arterial Stiffness Responses to Muscle Metaboreflex Activation With Concurrent Cold Pressor Test. Am J Hypertens. 2015 Nov;28(11):1332-8. doi: 10.1093/ajh/hpv043. Epub 2015 Apr 22. PMID 25904650